CLINICAL TRIAL: NCT02692703
Title: A Single-Arm, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of ABT-493/ABT-530 in Adult Post-Liver or Post-Renal Transplant Recipients With Chronic Hepatitis C Virus Genotype 1 - 6 Infection (MAGELLAN-2)
Brief Title: A Study to Evaluate the Safety and Efficacy of ABT-493/ABT-530 in Adult Post-Liver or Post-Renal Transplant Recipients With Chronic Hepatitis C Virus (MAGELLAN-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-596; 2015-005616-14 (EudraCT Number)
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; HCV; Hepatitis C Virus
Keywords: HCV Treatment Experienced; Hepatitis C; HCV Genotype 3; Without cirrhosis; Non-cirrhotic; HCV Genotype 2; Renal Transplant; HCV Treatment Naive; Post transplant; HCV Genotype 6; Liver Transplant; HCV Genotype 5; HCV Genotype 4; Kidney Transplant; HCV Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir and pibrentasvir; glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Glecaprevir/Pibrentasvir (Experimental): Glecaprevir/pibrentasvir (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: glecaprevir/pibrentasvir — Tablet; glecaprevir coformulated with pibrentasvir
  Other Names: glecaprevir also known as ABT-493; pibrentasvir also known as ABT-530; MAVYRET

SUMMARY:
The purpose of this study is to assess the safety and efficacy of 12 weeks of treatment of ABT-493/ABT-530 (glecaprevir/pibrentasvir) in adults who are post primary orthotopic liver or renal transplant with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at time of screening.
* Screening laboratory result indicating hepatitis C virus (HCV) genotype 1-6 (GT1-6) infection.
* Subject is a recipient of a cadaveric or living donor liver transplant which was a consequence of HCV infection at least 3 months prior to screening Or subject received a cadaveric or living donor kidney at least 3 months before screening.
* Subjects must be documented as non-cirrhotic.
* Subject is currently taking a stable immunosuppression regimen based on tacrolimus, sirolimus, everolimus, mycophenolate mofetil (MMF), mycophenolic acid, azathioprine, and/or cyclosporine.

Exclusion Criteria:

* Female subject who is pregnant, breastfeeding or is considering becoming pregnant during the study or for approximately 30 days after the last dose of study drug.
* Clinical history of fibrosing cholestatic hepatitis post-transplant.
* Re-transplantation of the liver or kidney.
* Steroid resistant rejection of the transplanted liver or kidney, or a history of rejection treated with high dose steroid within 3 months of screening.
* History of post-transplant complications related to hepatic or renal vasculature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rhee, MD, Study Director — AbbVie

REFERENCES:
- [Background] Reau N, Kwo PY, Rhee S, Brown RS Jr, Agarwal K, Angus P, Gane E, Kao JH, Mantry PS, Mutimer D, Reddy KR, Tran TT, Hu YB, Gulati A, Krishnan P, Dumas EO, Porcalla A, Shulman NS, Liu W, Samanta S, Trinh R, Forns X. Glecaprevir/Pibrentasvir Treatment in Liver or Kidney Transplant Patients With Hepatitis C Virus Infection. Hepatology. 2018 Oct;68(4):1298-1307. doi: 10.1002/hep.30046. Epub 2018 Jul 25. PMID 29672891
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 36-day screening period.
Period: Overall Study
Arm/Group | Glecaprevir/Pibrentasvir
Started | 100
Completed | 98
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.19 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 8
  White | 78
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority of the percentage of participants who achieved SVR12 compared with the historical SVR12 rate for the current standard of care regimens (sofosbuvir [SOF]/ledipasvir [LDV] + ribavirin [RBV] OR SOF + daclatasvir [DCV] + RBV). Participants with missing data after backward imputation were counted as non-responders.
Time Frame: 12 weeks after the last dose of study drug (up to 24 weeks)
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 100
percentage of participants | 98 [95.3 to 100.0]
Statistical Analysis 1: Comparison: Glecaprevir/Pibrentasvir; Based on a 2-sided significance level of 0.05 and an underlying rate of ≥96%, 90 participants provides >90% power to demonstrate noninferiority of the regimen to the historical rate for current standard of care regimens (SOF/LDV + RBV OR SOF + DCV + RBV) (94%) (based on the normal approximation of a single binomial proportion in a one-sample test for superiority); Test type: Non-Inferiority — The noninferiority of the rate of sustained virologic response at 12 weeks after treatment as compared with the historical rate for the current standard of care regimens (SOF/LDV + RBV or SOF + DCV + RBV) was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 86% to achieve noninferiority; Percentage of Participants = 98, 95% CI 2-sided [95.3 to 100.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Up to 12 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 100
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug (up to 12 weeks)
Population: All participants who received at least 1 dose of study drug, completed treatment, had HCV RNA <LLOQ at the final treatment visit, and had post-treatment data available, excluding reinfection.
Measure: Number; unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 99
percentage of participants | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 8/100
Other Adverse Events (participants affected / at risk) | 67/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=100)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1)
Immunosuppressant drug level increased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=100)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (11)
Nausea (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 5 (8)
Fatigue (General disorders) | 22 (26)
Upper respiratory tract infection (Infections and infestations) | 8 (10)
Urinary tract infection (Infections and infestations) | 5 (6)
Viral upper respiratory tract infection (Infections and infestations) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Dizziness (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 22 (26)
Insomnia (Psychiatric disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT02692703/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT02692703/SAP_001.pdf